CLINICAL TRIAL: NCT06395740
Title: Comparison Between Incidence of Pneumonia in Non-ventilated Cerebrovascular Stroke Patients Suffering from Bulbar Palsy Depending on Nasogastric Tube Feeding and Those Who Are Totally Parenterally Fed.
Brief Title: Aspiration Pneumonia in Cerebrovascular Stroke Patients Suffering from Bulbar Palsy
Acronym: TPN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMASU R65/2024
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-03

CONDITIONS: Aspiration Pneumonia
MeSH Terms: conditions — Pneumonia, Aspiration

STUDY DESIGN:
Intervention Model Description: All participants are to be resuscitated at first and second days of admission keeping all of them NPO then to be randomly divided according to the method of obtaining their nutritional needs into two groups. Energy target will be set at 30 kcal/ kg IBW in males and 25 Kcal/kg IBW in females, while protein requirements will be set at 1.2 g/kg IBW
  First group (group A):
  Group A patients will be scheduled for continuation of NPO strategy except for medications to be given via nasogastric tube till 14 days from day of stroke with fulfilment of nutrition requirement by parenteral route guided by Aspen2020 guidelines.
  Second group (group B):
  Group B patients will be scheduled for enteral nutrition via nasogastric tube.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- enteral nutrition group (Experimental): patients will be scheduled for enteral nutrition via nasogastric tube.The amount of nasogastric feed given each day will be calculated according to the patient's calorie requirement and administered as 100 ml nasogastric tube feeding every four hours escalating to 200 ml every four hours according to patients' toleration and caloric needs. Patients will be positioned at ≥ 45° head-end elevation during feeds. They will be observed regularly during feeds, and the position of the nasogastric tube will be confirmed before each feed by auscultation by stethoscope.
  Interventions: Other: Enteral nutrtion
- total parentral nutrition group (Experimental): patients will be scheduled for continuation of NPO strategy except for medications to be given via nasogastric tube till 14 days from day of stroke with fulfilment of nutrition requirement by parenteral route
  Interventions: Other: TPN

INTERVENTIONS:
Other: Enteral nutrtion — enteral nutrition via nasogastric tube.
  Arms: enteral nutrition group
Other: TPN — of NPO strategy except for medications to be given via nasogastric tube till 14 days from day of stroke with fulfilment of nutrition requirement by parenteral route
  Arms: total parentral nutrition group

SUMMARY:
One of the most serious complications in the critically ill patient complaining of bulbar palsy is aspiration pneumonia. These patients are scheduled for nasogastric tube feeding trying to avoid recurrent aspiration and subsequent aspiration pneumonia. Even though, the risk of aspiration is still present. Putting a total parenteral nutrition regimen for these patients is a supposed strategy to avoid aspiration pneumonia till recovery from bulbar palsy or planning for tracheostomy and or feeding gastrostomy.

DETAILED DESCRIPTION:
Aspiration pneumonia in cerebrovascular patients suffering from bulbar palsy can reach up to 60 %. (Martino R et al., 2012). All swallowing stages can be affected in cerebrovascular stroke patients. Difficulty in deglutition lower oesophageal sphincter dysfunction, delayed gastric empty and subsequent increase in gastric residual volume and decreased lower oesophageal sphincter tone and subsequent increase in gastroesophageal reflux all can be found in patients suffering from cerebrovascular stroke. (Schaller BJ et al., 2006).

As enteral feeding via oral route is risky in patients suffering from bulbar palsy, nasogastric tube is being used as a mode of enteral feeding till recovery from bulbar palsy or doing a gastrostomy tube as an alternative mode for enteral feeding. There is no survival benefit for early enteral feeding via nasogastric tube when compared with delayed tube feeding as formulated by the Feed or Ordinary Diet (FOOD) trial and suggested delaying nasogastric feeding may decrease mortality in bulbar palsy patients (Dennis MS et al., 2005).

Although this is the common practice to get the nutritional needs, there is evidence that early enteral feeding is not nutritionally superior to early TPN administration. Moreover, there is more rapid recovery of both albumin and protein in patients started TPN rather than those of enteral feeding at least for the first 2 weeks of stroke which is the time of maximum risk of malnutrition (Yamada SM, 2015).

Bulbar palsy non ventilated cerebrovascular patients who are scheduled for nasogastric tube feeding are at a high risk of aspiration pneumonia, with incidence from 33% to 70% (Langdon PC et al., 2009). Dysfunction of Lower oesophageal sphincter is exaggerated by nasogastric tube, that means increase of incidence of gastroesophageal reflux and micro aspiration (Gomes GF., 2003). Also, nasogastric tube can be colonized by gram negative bacteria as nasogastric tube change gastric acidity and promote bacterial colonization and increasing risk of micro aspiration and sequent aspiration pneumonia (Spilker CA et al., 1996). So non ventilated cerebrovascular stroke patients suffering from bulbar palsy and scheduled for nasogastric tube enteral feeding are at risk of aspiration pneumonia (Warusevitane A et al., 2014).

Even though parenteral feeding has the advantage of protection from aspiration pneumonia, it has risk of complications like hyperglycaemia, refeeding-syndrome, bone demineralisation, catheter infections), fortunately these complications can be minimised by carefully monitoring patients and the use of teams for nutrition support especially during long-term PN.( Hartl WH et al., 2009)

Our goal in this study is to compare the incidence of aspiration pneumonia when keeping patients on total parenteral feeding regimen in comparison with early start of enteral feeding with nasogastric tube during early stage of stroke in stroke patients suffering from bulbar palsy.

ELIGIBILITY:
Inclusion Criteria:

* 1. cerebrovascular stroke patients either ischemic or haemorrhagic within first 7 days 2. Age above 18 years 3. patients suffering from bulbar palsy.

Exclusion Criteria:

- Mechanically ventilated patients at first presentation. 2. Patients suffering from attacks of fits. 3. Patients suffering from signs and symptoms of pneumonia before attack of cerebrovascular stroke.

4. Patients suffering from degenerative neurological diseases. 5. Patients with developmental delay or neurological disease. 6. Patients with hepatic or renal coma. 7. Patients with hemodynamic instability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-05 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of pneumonia | within 14 days from inclusion in study
  guided by The British Thoracic Society recommendations for definition pneumonia

SECONDARY OUTCOMES:
mechanical ventilation | 30 days from inclusion in the study,
  Incidence of mechanical ventilation in both groups
mortality rate | 30 days from inclusion in the study,
  incidence of mortality in both groups
catheter related infection | 14 days from inclusion in study
  incidence of catheter related infection

CONTACTS AND LOCATIONS:
Overall Officials: Adel ELansary, Principal Investigator — Faculty of medicine, Ain Shams university
Locations (1):
- Abdallah Mahmoud Zaki Soudi, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: starting 6 months after publication